CLINICAL TRIAL: NCT06497985
Title: A Randomised, Open-label, Multicenter Phase III Study of Tucidinostat in Combination With Sintilimab and Bevacizumab in MSS/pMMR Colorectal Cancer Patients Who Failed at Least Second-line Standard Therapies
Brief Title: A Study of Tucidinostat in Combination With Sintilimab and Bevacizumab in MSS/pMMR Colorectal Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDM303
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; sintilimab; Bevacizumab; HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tucidinostat+sintilimab+bevacizumab (Experimental)
  Interventions: Drug: Tucidinostat; Drug: Sintilimab; Drug: Bevacizumab
- fruquintinib (Active Comparator)
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Tucidinostat — 30mg orally BIW
  Other Names: Chidamide
  Arms: tucidinostat+sintilimab+bevacizumab
Drug: Sintilimab — 200 mg intravenously (IV) Q3W
  Arms: tucidinostat+sintilimab+bevacizumab
Drug: Bevacizumab — 7.5mg/kg intravenously (IV) Q3W
  Arms: tucidinostat+sintilimab+bevacizumab
Drug: Fruquintinib — 5mg orally QD
  Arms: fruquintinib

SUMMARY:
A randomised, open-label, multicenter phase III study to evaluate the efficacy and safety of tucidinostat in combination with sintilimab and bevacizumab versus fruquintinib monotherapy in MSS/pMMR colorectal cancer patients.

DETAILED DESCRIPTION:
This is a randomised, open-label, multicenter phase III study evaluating the efficacy and safety of tucidinostat in combination with sintilimab and bevacizumab versus fruquintinib monotherapy in MSS/pMMR colorectal cancer patients. 430 patients will be randomised (1:1) to receive tucidinostat in combination with sintilimab and bevacizumab (experimental arm) or fruquintinib monotherapy (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent for the study.
2. Age ≥18 years and ≤75 years.
3. Histologically or cytologically confirmed unresectable and metastatic colorectal adenocarcinoma.
4. Has been previously treated and has shown disease progression or could not tolerate standard treatment, which must include fluoropyrimidine, irinotecan and oxaliplatin, with or without an anti-vascular endothelial growth factor (VEGF) monoclonal antibody (bevacizumab) or anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (cetuximab or panitumumab) .
5. Have confirmed MSS or MSI-L, or pMMR.
6. KRAS status must have been previously determined (mutant or wild-type) .
7. Measurable disease per RECIST v1.1.
8. ECOG PS 0 or 1.
9. Adequate organ function.
10. Expected survival >12 weeks.

Exclusion Criteria:

1. Prior use of HDAC inhibitor.
2. Received prior therapies targeting PD-1, PD-L1, CTLA4, or any other immune checkpoint pathway.
3. Prior use of small-molecule tyrosine kinase inhibitor of VEGF receptors.
4. Received any anti-tumor therapy or investigational agent and device within 28 days before the first dose of study treatment.
5. Received radiotherapy within 28 days before the first dose of study treatment.
6. If randomized into the control group, it is planned to use the combination of tucidinostat with PD-1 inhibitor and bevacizumab after the end of study treatment.
7. History of autoimmune diseases requiring systemic treatment within 2 years before the first dose of study treatment.
8. Known history of primary immunodeficiency.
9. Received systemic immunosuppressive drugs within 28 days before the first dose of study treatment.
10. Received systemic immunostimulatory drugs within 28 days before the first dose of study treatment.
11. Received major surgery within 28 days before the first dose of study treatment.
12. Received a live vaccine within 28 days before the first dose of study treatment or planned to receive during the study period.
13. Has not recovered ( ≤ Grade 1 defined by CTCAE V5.0) from AEs due to prior anti-cancer therapy.
14. Has uncontrolled diabetes assessed by investigators within 7 days before the first dose of study treatment.
15. Has symptomatic and untreated central nervous system (CNS) metastases.
16. Has uncontrollable or major cardiovascular disease.
17. History of cerebrovascular accidents within 6 months before the first dose of study treatment.
18. History of serious thromboembolism within 6 months before the first dose of study treatment.
19. History of gastrointestinal perforation and/or fistula etc., within 6 months before the first dose of study treatment.
20. Obvious gastrointestinal abnormalities during the screening period,which may affect the intake, transport or absorption of drugs.
21. Known history of bleeding disorders or coagulopathy.
22. Anticoagulants or thrombolytic agents are being used during the screening period.
23. Uncontrolled pleural/abdominal/pericardial effusion that was drained within 14 days before the first dose of study treatment.
24. Suspected interstitial lung disease (ILD) or pulmonary fibrosis or pulmonary inflammation requiring treatment.
25. Severe or active infection requiring systemic therapy.
26. Known active pulmonary tuberculosis.
27. Active hepatitis B or hepatitis C.
28. HIV positive or syphilis infection.
29. History of malignant tumor.
30. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
31. History of hypersensitivity to study drugs, or any of its excipients.
32. History of alcohol or drug abuse.
33. Unwilling or unable to comply with procedures required in this protocol.
34. Pregnant or breast-feeding women. Male/Female is unwilling or unable to use a highly effective method of birth control.
35. Any condition not suitable for participating in the trial in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  From randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS assessed by investigator per RECIST v1.1, measured from the date of randomization until progression or death, whichever occurs first.
Overall response rate (ORR) | Up to approximately 2 years
  Proportion of participants who achieved complete response (CR) or partial response (PR) assessed by investigator according to RECIST v1.1.
Duration of response (DOR) | Up to approximately 2 years
  From the first occurrence of PR or CR until the date of first documented progression according to RECIST 1.1, or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 2 years
  Proportion of participants who achieved CR or PR, or stable disease (SD) assessed by investigator according to RECIST v1.1.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life (QOL) Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life Scale Score | Up to approximately 2 years
  EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire, contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and global health status/QOL scale.Change from baseline in the EORTC QLQ-C30 Global Health Status/Quality of Life Scale scores will be presented.
Change From Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Health Utility Index Scores | Up to approximately 2 years
  The EQ-5D-5L is a self-reported health status questionnaire that consisted of 2 components: health state profile and optional VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: no problem, slight problem, moderate problem, severe problem, and extreme problem. Change from baseline in health utility index scores will be presented.
Change From Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS) Score | Up to approximately 2 years
  EQ-5D-5L consisted of 2 components: health state profile and optional VAS. The VAS records the respondent's self-rated health on a vertical visual analogue scale. The VAS 'thermometer' has endpoints of 100 (Best imaginable health state) at the top and 0 (Worst imaginable health state) at the bottom. Change from baseline in EQ-5D-5L VAS scores will be presented.
Safety and Tolerability | Up to approximately 2 years
  Number of Participants Who Experience an Adverse Event (AE) assessed by CTCAE v5.0.
Plasma concentrations of tucidinostat | Up to approximately 6 months
  Plasma samples were collected from the participants at the defined time points. Plasma concentrations were measured using a validated, specific, and sensitive method.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Rui-Hua Xu, Guangzhou, Guangdong, China